CLINICAL TRIAL: NCT04045457
Title: A Study to Determine the Tissue Properties, Vascular Physiology and Biochemical Milieu of Myofascial Trigger Points
Acronym: MTrP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Naomi Lynn Gerber, Professor, George Mason University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PR00005701; R01AR057348 (NIH)
Record Dates: First submitted 2016-06-10; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Myofascial Pain
Keywords: active trigger points
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIngle arm (Other): Single arm, intervention All recipients were treated with dry needling technique into active myofascial trigger points They received 1 treatment weekly for three weeks.
  Interventions: Procedure: dry needling

INTERVENTIONS:
Procedure: dry needling — insertion of needle into active myofascial trigger point

SUMMARY:
Determine the effect of dry needling using a 32 gauge needle on active trigger points in subjects with chronic myofascial pain.

Participants will receive treatment for active trigger points (3 on successive weeks) and will have pain, status of the trigger point and functional measures assessed at baseline, after treatment and eight weeks later.

DETAILED DESCRIPTION:
Chronic myofascial pain syndromes, such as pain associated with myofascial trigger points (MTrPs), are prevalent yet poorly understood. Our long-term goal is to determine the pathogenesis and pathophysiological mechanisms of chronic pain associated with trigger points, eventually leading to the development of objective diagnostic criteria and effective pain management strategies. We propose to achieve this goal using a new and unique integrative methodology combining microanalytic biochemical assays, ultrasound technology (imaging) and mathematical modeling. An additional component of the study plan is to learn if a standard treatment for MTrPs is associated with the biochemical and ultrasound changes we will be measuring This project has the following specific aims: 1) To understand the viscoelastic soft tissue neighborhood and vascular physiology of affected muscle at a macroscopic level using ultrasound imaging, elastography and Doppler blood flow imaging; 2) To understand the pathophysiology of myofascial trigger points at a nanotechnological level through assays of biochemical milieu using a microdialysis technique; 3) To develop mathematical models of underlying pathophysiological mechanisms based on experimental observations for quantitative hypothesis testing; 4) To determine if dry needle therapy, a standard of care for MTrPs, changes the macroscopic and/or microscopic measurements and leads to resolution of the trigger point and secondarily associated pain symptoms.. Our hypothesis is that pathogenesis of myofascial pain syndrome involves local trauma to the muscle fibers, and the biochemical response to the injury leads to sustained muscle contracture, compression of blood vessels and a local energy crisis that causes tissue hypoxia and the expression of pain-producing substances at myofascial trigger points. Relieving the trigger point through dry needle therapy

ELIGIBILITY:
Inclusion Criteria:

* spontaneous soft tissue pain in shoulder and neck region

Exclusion Criteria:

* recent fracture, neurological injury or history of stroke, use of opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Verbal Analog Scale | change from baseline to 3 weeks and at 8 weeks
  scale of 0-10 as a measure of pain severity
Presence of myofascial trigger point | change from baseline to 3 weeks and at 8 weeks
  Digital palpation of the trigger point was performed by investigators and scored as present or absent; if present was it associated with spontaneous pain or was pain induced with palpation
Brief Pain Inventory | change from baseline to 3 weeks and at 8 weeks
  Validated scale of pain severity and interference

SECONDARY OUTCOMES:
Oswestry Disability Scale | change from baseline to 3 weeks and at 8 weeks
  self-reports of disability
MOS-short form 36 v2 | change from baseline to 3 weeks and at 8 weeks
  self-reports of disability and health related quality of life Profile of Mood States, range of motion of neck and shoulder, manual muscle test)
Manual Muscle test | change from baseline to 3 weeks and at 8 weeks
  grade strength 0-5, neck and shoulder girdle muscle
Profile of Mood States | change from baseline to 3 weeks and at 8 weeks
  measures of mood and affect (depression and anxiety)
range of motion | change from baseline to 3 weeks and at 8 weeks
  shoulder and neck range of motion in degrees

REFERENCES:
- [Result] Turo D, Otto P, Hossain M, Gebreab T, Armstrong K, Rosenberger WF, Shao H, Shah JP, Gerber LH, Sikdar S. Novel Use of Ultrasound Elastography to Quantify Muscle Tissue Changes After Dry Needling of Myofascial Trigger Points in Patients With Chronic Myofascial Pain. J Ultrasound Med. 2015 Dec;34(12):2149-61. doi: 10.7863/ultra.14.08033. Epub 2015 Oct 21. PMID 26491094
- [Result] Gerber LH, Shah J, Rosenberger W, Armstrong K, Turo D, Otto P, Heimur J, Thaker N, Sikdar S. Dry Needling Alters Trigger Points in the Upper Trapezius Muscle and Reduces Pain in Subjects With Chronic Myofascial Pain. PM R. 2015 Jul;7(7):711-718. doi: 10.1016/j.pmrj.2015.01.020. Epub 2015 Feb 4. PMID 25661462
- [Result] Gerber LH, Sikdar S, Armstrong K, Diao G, Heimur J, Kopecky J, Turo D, Otto P, Gebreab T, Shah J. A systematic comparison between subjects with no pain and pain associated with active myofascial trigger points. PM R. 2013 Nov;5(11):931-8. doi: 10.1016/j.pmrj.2013.06.006. Epub 2013 Jun 28. PMID 23810811
- [Result] Turo D, Otto P, Shah JP, Heimur J, Gebreab T, Zaazhoa M, Armstrong K, Gerber LH, Sikdar S. Ultrasonic characterization of the upper trapezius muscle in patients with chronic neck pain. Ultrason Imaging. 2013 Apr;35(2):173-87. doi: 10.1177/0161734612472408. PMID 23493615